CLINICAL TRIAL: NCT03834194
Title: Effect of Incentives for Self-weighing, Weight Management Goals and Physical Activity Goals on Gaining Weight Healthily During Pregnancy
Brief Title: Gestational Weight and Incentive Research Study
Acronym: Bloom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-06293-XP
Record Dates: First submitted 2019-01-03; First posted 2019-02-07 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2020-03

CONDITIONS: Gestational Weight Gain
Keywords: excessive weight gain; pregnancy
MeSH Terms: conditions — Gestational Weight Gain | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Lottery + Monthly Weight (Experimental): Participants will be eligible for a daily lottery if they have weighed themselves in the previous day on the e-scale. For each day of the study, participants will be informed of the study's randomly-generated winning lottery number and their winnings ($0, $2, $15 or not eligible for lottery due to lack of weighing). Participants will receive $14 per month if they have gained within the recommended monthly range for their BMI category. Otherwise, participants will be specifically notified that they would have received $14 had they had gained within the recommended range for the month, drawing on research showing that loss aversion can be motivating.
  Interventions: Behavioral: Lottery + Monthly Weight
- Lottery + Overall Weight + Exercise (Experimental): Participants will be eligible for a daily lottery if they have weighed themselves in the previous day on the e-scale. For each day of the study, participants will be informed of the study's randomly-generated winning lottery number and their winnings if any. Participants will be given the IOM GWG recommendation based on their body mass index at randomization, adjusted for data collection at 36 weeks. If they achieve the goal at 36 weeks, they will receive $112 after the data collection visit. Participants will be asked to engage in 150 minutes of exercise each week based on the guideline from the ACOG. They will receive $3.50 if they meet their activity goal for the week. Otherwise, they will be notified that they would have received $3.50 had they meet their activity goal.
  Interventions: Behavioral: Lottery + Overall Weight + Exercise
- Lottery + Overall Weight (Experimental): Participants will be eligible for a daily lottery if they have weighed themselves in the previous day on the e-scale. For each day of the study, participants will be informed of the study's randomly-generated winning lottery number and their winnings ($0, $2, $15 or not eligible for lottery due to lack of weighing). Participants will be given the Institute of Medicine gestational weight gain recommendation based on their body mass index at randomization, adjusted for data collection at 36 weeks. If they achieve the goal at 36 weeks, they will receive $112 after the data collection visit.
  Interventions: Behavioral: Lottery + Overall Weight
- Lottery + Monthly Weight + Exercise (Experimental): Participants will be eligible for a daily lottery if they have weighed themselves in the previous day on the e-scale. For each day of the study, participants will be informed of the study's randomly-generated winning lottery number and their winnings if any. Participants will receive $14 per month if they have gained within the recommended monthly range for their BMI category. Otherwise, they will be notified that they would have received $14 had they had gained within the recommendation for the month. Participants will be asked to engage in 150 minutes of exercise each week based on the guideline from the ACOG. They will receive $3.50 if they meet their activity goal for the week. Otherwise, they will be notified that they would have received $3.50 had they meet their activity goal.
  Interventions: Behavioral: Lottery + Monthly Weight + Exercise
- Loss + Monthly Weight (Experimental): Participants randomized to an arm that contains the self-weighing (certain loss) component will have a balance of $3.50 at the beginning of each week of the the study and each day that they do not weigh, $0.50 will be subtracted from this account. Participants will receive $14 per month if they have gained within the recommended monthly range for their BMI category. Otherwise, participants will be specifically notified that they would have received $14 had they had gained within the recommended range for the month, drawing on research showing that loss aversion can be motivating.
  Interventions: Behavioral: Loss + Monthly Weight
- Loss + Overall Weight + Exercise (Experimental): Participants randomized to an arm that contains the self-weighing (certain loss) component will have a balance of $3.50 at the beginning of each week of the study and each day that they do not weigh, $0.50 will be subtracted from this account. Participants will be given the IOM GWG recommendation based on their body mass index at randomization, adjusted for data collection at 36 weeks. If they achieve the goal at 36 weeks, they will receive $112 after the data collection visit. Participants will be asked to engage in 150 minutes of exercise each week based on the guideline from the ACOG. They will receive $3.50 if they meet their activity goal for the week. Otherwise, they will be notified that they would have received $3.50 had they meet their activity goal.
  Interventions: Behavioral: Loss + Overall Weight + Exercise
- Loss + Overall Weight (Experimental): Participants randomized to an arm that contains the self-weighing (certain loss) component will have a balance of $3.50 at the beginning of each week of the the study and each day that they do not weigh, $0.50 will be subtracted from this account. Participants will be given the Institute of Medicine gestational weight gain recommendation based on their body mass index at randomization, adjusted for data collection at 36 weeks. If they achieve the goal at 36 weeks, they will receive $112 after the data collection visit.
  Interventions: Behavioral: Loss + Overall Weight
- Loss + Monthly Weight + Exercise (Experimental): Participants randomized to an arm that contains the self-weighing (certain loss) component will have a balance of $3.50 at the beginning of each week of the study and each day that they do not weigh, $0.50 will be subtracted from this account. Participants will receive $14 per month if they have gained within the recommended monthly range for their BMI category. Otherwise, they will be notified that they would have received $14 had they had gained within the recommendation for the month. Participants will be asked to engage in 150 minutes of exercise each week based on the guideline from the ACOG. They will receive $3.50 if they meet their activity goal for the week. Otherwise, they will be notified that they would have received $3.50 had they meet their activity goal.
  Interventions: Behavioral: Loss + Monthly Weight + Exercise

INTERVENTIONS:
Behavioral: Lottery + Monthly Weight — Lottery for daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) on a monthly basis.
  Arms: Lottery + Monthly Weight
Behavioral: Lottery + Overall Weight + Exercise — Lottery for daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) by the end of the study.
  Incentives for meeting an exercise goal of 150 minutes of moderate physical activity per week, as recommended by the American College of Obstetricians and Gynecologists.
  Arms: Lottery + Overall Weight + Exercise
Behavioral: Lottery + Overall Weight — Lottery for daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) by the end of the study.
  Arms: Lottery + Overall Weight
Behavioral: Loss + Overall Weight — Certain loss for not engaging in daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) by the end of the study.
  Arms: Loss + Overall Weight
Behavioral: Loss + Overall Weight + Exercise — Certain loss for not engaging in daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) by the end of the study.
  Incentives for meeting an exercise goal of 150 minutes of moderate physical activity per week, as recommended by the American College of Obstetricians and Gynecologists.
  Arms: Loss + Overall Weight + Exercise
Behavioral: Lottery + Monthly Weight + Exercise — Lottery for daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) on a monthly basis.
  Incentives for meeting an exercise goal of 150 minutes of moderate physical activity per week, as recommended by the American College of Obstetricians and Gynecologists.
  Arms: Lottery + Monthly Weight + Exercise
Behavioral: Loss + Monthly Weight — Certain loss for not engaging in daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) on a monthly basis.
  Arms: Loss + Monthly Weight
Behavioral: Loss + Monthly Weight + Exercise — Certain loss for not engaging in daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) on a monthly basis.
  Incentives for meeting an exercise goal of 150 minutes of moderate physical activity per week, as recommended by the American College of Obstetricians and Gynecologists.
  Arms: Loss + Monthly Weight + Exercise

SUMMARY:
Bloom is a research study that examines whether incentives for daily self-weighing, weekly physical activity, monthly weight management or overall (from enrollment up to 36 weeks pregnancy) weight management could help pregnant mothers manage a health weight gain during pregnancy.

DETAILED DESCRIPTION:
Gestational weight gain (GWG) is a serious public health concern, and 37% of normal weight, 64% of overweight, and 49-64% of obese women exceed the Institute of Medicine's GWG guidelines. [Deputy 2015] Excessive GWG increases the risk for illnesses, such as gestational diabetes mellitus (GDM) [Cheng 2008, Tovar 2009] which has a long-term impact on the health of both the mother (i.e., increased likelihood of developing metabolic syndrome, [Vohr 2008] type 2 diabetes, [Vambergue 2007, Bellamy 2009] and GDM in subsequent pregnancies [Bottalico 2007] and child [Vohr 2008].

For weight loss, research has found that modest financial incentives are a promising pragmatic strategy for an intervention. Yet, most previous weight management research that has utilized incentives has targeted weight outcomes rather than the behaviors necessary to achieve them. [Paul-Ebhohimhen 2008, Burns 2012] For self-weighing, research has found that daily self-weighing is an important component that supplements behavioral interventions' effort in monitoring and managing gestational weight. [Phelan 2011, Olson 2017, Harrison 2013, Harrison 2014] For physical activity, research has found that physical activity may successfully manage GWG, and a greater adherence to the exercise program is linked to interventions that resulted in weight management success. [McDonald 2016] Thus, a strategy to increase adherence, like financial incentives, may be beneficial.

Consistent with recent research, [Leahey 2015] the investigators will incentivize daily self-weighing and participation in physical activity (i.e., the behaviors) in addition to GWG within the guidelines (i.e., the outcome). Behaviors that negatively impact health often involve immediate benefits and delayed costs (i.e., "eating for two" provides immediate gratification but may lead to excessive GWG), and many interventions involve immediate costs (i.e., the inconvenience and time of an intervention) with delayed and often uncertain benefits of better health years later. [Volpp 2011] Researchers also hypothesize that an approach that offers frequent chances to win small lotteries based on meeting short-term goals will be more effective than a straight pay-for-performance approach (of equal expected value) because people are emotionally attracted to the possibility of winning a lottery. [Loewenstein 2007, Volpp 2008] Therefore, the current study proposes to examine the impact of frequent chances to win small, proximal incentives for meeting short-term goals of self-weighing and physical activity and larger incentives for meeting overall GWG goals by the end of the 36-week gestational period.

To our knowledge, the study is the first to use financial incentives to reduce the likelihood of excessive GWG. This project will support evaluation of the feasibility of this promising approach to decreasing excessive GWG. The incentive strategy is based in theory and focuses on behaviors that has a strong link with gestational weight management (i.e., self-weighing and physical activity) and on an outcome (i.e., achievement of GWG goals), thereby moving the field forward in identifying promising approaches to incorporating financial incentives into gestational weight management. The study design is also pragmatic and has a strong potential for scalability and sustainability within the health care setting.

Pregnant participants (N=40) in their first trimester at an obstetric clinic in Memphis, TN will be randomized in a factorial experiment. Three intervention components will be randomized using a 2 x 2 x 2 factorial design: 1) daily incentives for self-weighing on an electronic scale that will transmit data to the study team (lottery/certain loss), 2) incentives for adhering to the Institute of Medicine's gestational weight gain guidelines based on BMI category (monthly/overall), and 3) incentives for reaching physical activity goals to manage gestational weight gain (yes/no).

Potential participants will be identified by the clinics' health professionals (i.e., nurses, obstetricians) at their pregnancy confirmation visit or will be self-identified through recruitment materials posted in the obstetric clinic (e.g., exam rooms, lobby and bathrooms). They will encouraged to contact the study team if they wish to learn more about the study and potentially enroll in the study. Upon recruitment, individuals who are interested in learning more about the study will be directed to the Way to Health web portal. Upon reaching the portal, potential participants will be asked to create an account and will then be informed of the details of the study, including its objectives, duration, requirements, and financial payments. If participants are still interested in participating, the Way to Health portal will take them through an automated online informed consent. Potential participants who click a clearly delineated button stating that they agree to participate in the study will be considered to have consented to enroll. After consenting, participants will complete an online questionnaire to determine their eligibility. Eligible participants will first answer a few questions about the number of pregnancies they have prior to the current one, age, annual household income, marital status, employment status, household size, education level, race, and ethnicity. Then, they will be randomized to one of the study arms and led through an automated description of the details specific to that arm. Participants will be provided with details regarding how to contact the research team via email or phone at any time if they subsequently wish to withdraw from the study. This contact information will remain easily accessible via the participants' individual Way to Health web portal dashboards throughout the study.

Participants will be randomized to one of 8 conditions, with combinations of 3 different components of incentive for GWG management and physical activity. Participants will be asked to complete daily self-weighing using the scale provided by the study, as well as wear a physical activity tracker.

Participants randomized to an arm that contains the self-weighing (lottery) component will be asked to pick a number between 00 and 99 at randomization, and will be informed that there will be a daily lottery, for which they will be eligible if they have weighed themselves in the previous day on the Withings e-scale. Then, for each day of their pregnancy, participants will be informed of the study's randomly-generated winning lottery number. Participants will be notified about the results of the lottery.

Participants randomized to an arm that contains the self-weighing (certain loss) component will have a portion of their incentives deducted from a weekly total.

Participants randomized to an arm that contains the monthly GWG incentive component will receive incentives for each month that they have gained within the recommended monthly range for their BMI category for the full months they are enrolled.

Participants randomized to an arm that contains the overall GWG incentive component will receive incentives for weight gain within the recommended range according to the Institute of Medicine gestational weight gain recommendation (based on their body mass index at randomization, adjusted for data collection at 36 weeks).

Participants randomized to an arm that contains the physical activity component will receive a weekly incentive if they achieved a 150 minute physical activity goal for each week based on the guideline from the American College of Obstetricians and Gynecologists (ACOG) [The American College of Obstetricians and Gynecologists 2015].

Measures will be obtained by trained research staff who are blinded to treatment assignment and who will be located within the obstetric clinic.

Baseline measures will be obtained in the first trimester. In-person follow-up data collection visits will be scheduled at gestational week 32 and week 36 (for those still pregnant at 36 weeks). Incentives ($30 for each follow-up visit) will be used to obtain high retention at all follow-up data collection visits. In addition, the research staff will attempt to schedule the data collection visits before or after regular office visits, in order to facilitate retention.

Weekly study meetings, which include retention as a standing agenda item, are also a component of this systematic and comprehensive approach. However, as the investigators will be recruiting participants at <12 weeks gestation (and miscarriage rates are highest in the first trimester), the investigators may lose up to 15% of participants due to miscarriage. [The American College of Obstetricians and Gynecologists 2015] Thus, the investigators project 20% attrition at the final data collection point (36 weeks gestation).

As this is a novel intervention, no related data exist to inform the effect size that might be expected, and as a pilot study, the trial is not powered to detect a significant difference between conditions.

Analyses of GWG (in kg) will be performed using mixed model longitudinal methods. Analyses of the proportion of women with excessive GWG will use logistic regression models to estimate the odds of an intervention participant's GWG falling below or above the guidelines, relative to staying within the recommendations. All of these analyses will inform effect size estimation for the full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* no greater than 12 weeks gestation upon recruitment (based on the date of their last menstrual period)
* have regular access to Wi-Fi or Bluetooth

Exclusion criteria:

* Greater than 12 week gestation up on recruitment (based on the health care provider's assessment)
* Underweight (BMI < 18.5) at baseline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Krukowski, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
IPD are protected by the Institutional Review Board (IRB) at the University of Tennessee Health Science Center (UTHSC). No individual without the IRB of UTHSC will have access to IDP.

REFERENCES:
- [Background] Deputy NP, Sharma AJ, Kim SY, Hinkle SN. Prevalence and characteristics associated with gestational weight gain adequacy. Obstet Gynecol. 2015 Apr;125(4):773-781. doi: 10.1097/AOG.0000000000000739. PMID 25751216
- [Background] Cheng YW, Chung JH, Kurbisch-Block I, Inturrisi M, Shafer S, Caughey AB. Gestational weight gain and gestational diabetes mellitus: perinatal outcomes. Obstet Gynecol. 2008 Nov;112(5):1015-22. doi: 10.1097/AOG.0b013e31818b5dd9. PMID 18978100
- [Background] Tovar A, Must A, Bermudez OI, Hyatt RR, Chasan-Taber L. The impact of gestational weight gain and diet on abnormal glucose tolerance during pregnancy in Hispanic women. Matern Child Health J. 2009 Jul;13(4):520-30. doi: 10.1007/s10995-008-0381-x. Epub 2008 Jul 3. PMID 18597166
- [Background] Vohr BR, Boney CM. Gestational diabetes: the forerunner for the development of maternal and childhood obesity and metabolic syndrome? J Matern Fetal Neonatal Med. 2008 Mar;21(3):149-57. doi: 10.1080/14767050801929430. PMID 18297569
- [Background] Vambergue A, Dognin C, Boulogne A, Rejou MC, Biausque S, Fontaine P. Increasing incidence of abnormal glucose tolerance in women with prior abnormal glucose tolerance during pregnancy: DIAGEST 2 study. Diabet Med. 2008 Jan;25(1):58-64. doi: 10.1111/j.1464-5491.2007.02306.x. Epub 2007 Nov 19. PMID 18028442
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams D. Type 2 diabetes mellitus after gestational diabetes: a systematic review and meta-analysis. Lancet. 2009 May 23;373(9677):1773-9. doi: 10.1016/S0140-6736(09)60731-5. PMID 19465232
- [Background] Bottalico JN. Recurrent gestational diabetes: risk factors, diagnosis, management, and implications. Semin Perinatol. 2007 Jun;31(3):176-84. doi: 10.1053/j.semperi.2007.03.006. PMID 17531899
- [Background] Paul-Ebhohimhen V, Avenell A. Systematic review of the use of financial incentives in treatments for obesity and overweight. Obes Rev. 2008 Jul;9(4):355-67. doi: 10.1111/j.1467-789X.2007.00409.x. Epub 2007 Oct 23. PMID 17956546
- [Background] Burns RJ, Donovan AS, Ackermann RT, Finch EA, Rothman AJ, Jeffery RW. A theoretically grounded systematic review of material incentives for weight loss: implications for interventions. Ann Behav Med. 2012 Dec;44(3):375-88. doi: 10.1007/s12160-012-9403-4. PMID 22907712
- [Background] Phelan S, Jankovitz K, Hagobian T, Abrams B. Reducing excessive gestational weight gain: lessons from the weight control literature and avenues for future research. Womens Health (Lond). 2011 Nov;7(6):641-61. doi: 10.2217/whe.11.70. PMID 22040207
- [Background] Olson CM, Strawderman MS, Graham ML. Association between consistent weight gain tracking and gestational weight gain: Secondary analysis of a randomized trial. Obesity (Silver Spring). 2017 Jul;25(7):1217-1227. doi: 10.1002/oby.21873. Epub 2017 Jun 2. PMID 28573669
- [Background] Harrison CL, Lombard CB, Strauss BJ, Teede HJ. Optimizing healthy gestational weight gain in women at high risk of gestational diabetes: a randomized controlled trial. Obesity (Silver Spring). 2013 May;21(5):904-9. doi: 10.1002/oby.20163. PMID 23784892
- [Background] Harrison CL, Teede HJ, Lombard CB. How effective is self-weighing in the setting of a lifestyle intervention to reduce gestational weight gain and postpartum weight retention? Aust N Z J Obstet Gynaecol. 2014 Aug;54(4):382-5. doi: 10.1111/ajo.12207. Epub 2014 Apr 16. PMID 24738837
- [Background] McDonald SM, Liu J, Wilcox S, Lau EY, Archer E. Does dose matter in reducing gestational weight gain in exercise interventions? A systematic review of literature. J Sci Med Sport. 2016 Apr;19(4):323-35. doi: 10.1016/j.jsams.2015.03.004. Epub 2015 Mar 26. PMID 25846125
- [Background] Leahey TM, Subak LL, Fava J, Schembri M, Thomas G, Xu X, Krupel K, Kent K, Boguszewski K, Kumar R, Weinberg B, Wing R. Benefits of adding small financial incentives or optional group meetings to a web-based statewide obesity initiative. Obesity (Silver Spring). 2015 Jan;23(1):70-6. doi: 10.1002/oby.20937. Epub 2014 Nov 11. PMID 25384463
- [Background] Volpp KG, Asch DA, Galvin R, Loewenstein G. Redesigning employee health incentives--lessons from behavioral economics. N Engl J Med. 2011 Aug 4;365(5):388-90. doi: 10.1056/NEJMp1105966. No abstract available. PMID 21812669
- [Background] Loewenstein G, Brennan T, Volpp KG. Asymmetric paternalism to improve health behaviors. JAMA. 2007 Nov 28;298(20):2415-7. doi: 10.1001/jama.298.20.2415. No abstract available. PMID 18042920
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Gardner B, Wardle J, Poston L, Croker H. Changing diet and physical activity to reduce gestational weight gain: a meta-analysis. Obes Rev. 2011 Jul;12(7):e602-20. doi: 10.1111/j.1467-789X.2011.00884.x. Epub 2011 Apr 27. PMID 21521451
- [Background] Oken E, Taveras EM, Kleinman KP, Rich-Edwards JW, Gillman MW. Gestational weight gain and child adiposity at age 3 years. Am J Obstet Gynecol. 2007 Apr;196(4):322.e1-8. doi: 10.1016/j.ajog.2006.11.027. PMID 17403405
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Mathews TJ. Births: final data for 2011. Natl Vital Stat Rep. 2013 Jun 28;62(1):1-69, 72. PMID 24974591
- [Background] Finkelstein EA, Linnan LA, Tate DF, Birken BE. A pilot study testing the effect of different levels of financial incentives on weight loss among overweight employees. J Occup Environ Med. 2007 Sep;49(9):981-9. doi: 10.1097/JOM.0b013e31813c6dcb. PMID 17848854
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] Yancy WS Jr, Shaw PA, Wesby L, Hilbert V, Yang L, Zhu J, Troxel A, Huffman D, Foster GD, Wojtanowski AC, Volpp KG. Financial incentive strategies for maintenance of weight loss: results from an internet-based randomized controlled trial. Nutr Diabetes. 2018 May 25;8(1):33. doi: 10.1038/s41387-018-0036-y. PMID 29795365
- [Background] Shaw PA, Yancy WS Jr, Wesby L, Ulrich V, Troxel AB, Huffman D, Foster GD, Volpp K. The design and conduct of Keep It Off: An online randomized trial of financial incentives for weight-loss maintenance. Clin Trials. 2017 Feb;14(1):29-36. doi: 10.1177/1740774516669679. Epub 2016 Sep 23. PMID 27646508
- [Background] Patel MS, Asch DA, Troxel AB, Fletcher M, Osman-Koss R, Brady J, Wesby L, Hilbert V, Zhu J, Wang W, Volpp KG. Premium-Based Financial Incentives Did Not Promote Workplace Weight Loss In A 2013-15 Study. Health Aff (Millwood). 2016 Jan;35(1):71-9. doi: 10.1377/hlthaff.2015.0945. PMID 26733703
- [Background] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Heuer J, Sproat S, Hyson C, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults: A Randomized, Controlled Trial. Ann Intern Med. 2016 Mar 15;164(6):385-94. doi: 10.7326/M15-1635. Epub 2016 Feb 16. PMID 26881417
- [Derived] Krukowski R, Johnson B, Kim H, Sen S, Homsi R. A Pragmatic Intervention Using Financial Incentives for Pregnancy Weight Management: Feasibility Randomized Controlled Trial. JMIR Form Res. 2021 Dec 24;5(12):e30578. doi: 10.2196/30578. PMID 34951594
- See also: Tennessee Pregnancy Risk Assessment Monitoring System 2011 — https://www.tn.gov/content/dam/tn/health/documents/2011_TN_PRAMS_Summary_Report.pdf
- See also: The American College of Obstetricians and Gynecologists. Physical Activity and Exercise During Pregnancy and Postpartum Period. 2015 — https://www.acog.org/-/media/Committee-Opinions/Committee-on-Obstetric-Practice/co650.pdf?dmc=1&ts=20181004T1434361881
- See also: American College of Obstetricians and Gynecologists. Frequently Asked Questions (FAQ090). 2013 — https://www.acog.org/-/media/For-Patients/faq090.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Lottery + Monthly Weight: Participants will be eligible for a daily lottery if they have weighed themselves in the previous day on the e-scale. For each day of the study, participants will be informed of the study's randomly-generated winning lottery number and their winnings ($0, $2, $15 or not eligible for lottery due to lack of weighing). Participants will receive $14 per month if they have gained within the recommended monthly range for their BMI category. Otherwise, participants will be specifically notified that they would have received $14 had they had gained within the recommended range for the month, drawing on research showing that loss aversion can be motivating.
  Lottery + Monthly Weight: Lottery for daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) on a monthly basis.
- Lottery + Overall Weight + Exercise: Participants will be eligible for a daily lottery if they have weighed themselves in the previous day on the e-scale. For each day of the study, participants will be informed of the study's randomly-generated winning lottery number and their winnings if any. Participants will be given the IOM GWG recommendation based on their body mass index at randomization, adjusted for data collection at 36 weeks. If they achieve the goal at 36 weeks, they will receive $112 after the data collection visit. Participants will be asked to engage in 150 minutes of exercise each week based on the guideline from the ACOG. They will receive $3.50 if they meet their activity goal for the week. Otherwise, they will be notified that they would have received $3.50 had they meet their activity goal.
  Lottery + Overall Weight + Exercise: Lottery for daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) by the end of the study.
  Incentives for meeting an exercise goal of 150 minutes of moderate physical activity per week, as recommended by the American College of Obstetricians and Gynecologists.
- Lottery + Overall Weight: Participants will be eligible for a daily lottery if they have weighed themselves in the previous day on the e-scale. For each day of the study, participants will be informed of the study's randomly-generated winning lottery number and their winnings ($0, $2, $15 or not eligible for lottery due to lack of weighing). Participants will be given the Institute of Medicine gestational weight gain recommendation based on their body mass index at randomization, adjusted for data collection at 36 weeks. If they achieve the goal at 36 weeks, they will receive $112 after the data collection visit.
  Lottery + Overall Weight: Lottery for daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) by the end of the study.
- Lottery + Monthly Weight + Exercise: Participants will be eligible for a daily lottery if they have weighed themselves in the previous day on the e-scale. For each day of the study, participants will be informed of the study's randomly-generated winning lottery number and their winnings if any. Participants will receive $14 per month if they have gained within the recommended monthly range for their BMI category. Otherwise, they will be notified that they would have received $14 had they had gained within the recommendation for the month. Participants will be asked to engage in 150 minutes of exercise each week based on the guideline from the ACOG. They will receive $3.50 if they meet their activity goal for the week. Otherwise, they will be notified that they would have received $3.50 had they meet their activity goal.
  Lottery + Monthly Weight + Exercise: Lottery for daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) on a monthly basis.
  Incentives for meeting an exercise goal of 150 minutes of moderate physical activity per week, as recommended by the American College of Obstetricians and Gynecologists.
- Loss + Monthly Weight: Participants randomized to an arm that contains the self-weighing (certain loss) component will have a balance of $3.50 at the beginning of each week of the the study and each day that they do not weigh, $0.50 will be subtracted from this account. Participants will receive $14 per month if they have gained within the recommended monthly range for their BMI category. Otherwise, participants will be specifically notified that they would have received $14 had they had gained within the recommended range for the month, drawing on research showing that loss aversion can be motivating.
  Loss + Monthly Weight: Certain loss for not engaging in daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) on a monthly basis.
- Loss + Overall Weight + Exercise: Participants randomized to an arm that contains the self-weighing (certain loss) component will have a balance of $3.50 at the beginning of each week of the study and each day that they do not weigh, $0.50 will be subtracted from this account. Participants will be given the IOM GWG recommendation based on their body mass index at randomization, adjusted for data collection at 36 weeks. If they achieve the goal at 36 weeks, they will receive $112 after the data collection visit. Participants will be asked to engage in 150 minutes of exercise each week based on the guideline from the ACOG. They will receive $3.50 if they meet their activity goal for the week. Otherwise, they will be notified that they would have received $3.50 had they meet their activity goal.
  Loss + Overall Weight + Exercise: Certain loss for not engaging in daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) by the end of the study.
  Incentives for meeting an exercise goal of 150 minutes of moderate physical activity per week, as recommended by the American College of Obstetricians and Gynecologists.
- Loss + Overall Weight: Participants randomized to an arm that contains the self-weighing (certain loss) component will have a balance of $3.50 at the beginning of each week of the the study and each day that they do not weigh, $0.50 will be subtracted from this account. Participants will be given the Institute of Medicine gestational weight gain recommendation based on their body mass index at randomization, adjusted for data collection at 36 weeks. If they achieve the goal at 36 weeks, they will receive $112 after the data collection visit.
  Loss + Overall Weight: Certain loss for not engaging in daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) by the end of the study.
- Loss + Monthly Weight + Exercise: Participants randomized to an arm that contains the self-weighing (certain loss) component will have a balance of $3.50 at the beginning of each week of the study and each day that they do not weigh, $0.50 will be subtracted from this account. Participants will receive $14 per month if they have gained within the recommended monthly range for their BMI category. Otherwise, they will be notified that they would have received $14 had they had gained within the recommendation for the month. Participants will be asked to engage in 150 minutes of exercise each week based on the guideline from the ACOG. They will receive $3.50 if they meet their activity goal for the week. Otherwise, they will be notified that they would have received $3.50 had they meet their activity goal.
  Loss + Monthly Weight + Exercise: Certain loss for not engaging in daily self-weighing.
  Incentives for gaining weight within a recommended (by Institute of Medicine) on a monthly basis.
  Incentives for meeting an exercise goal of 150 minutes of moderate physical activity per week, as recommended by the American College of Obstetricians and Gynecologists.
Period: Overall Study
Arm/Group | Lottery + Monthly Weight | Lottery + Overall Weight + Exercise | Lottery + Overall Weight | Lottery + Monthly Weight + Exercise | Loss + Monthly Weight | Loss + Overall Weight + Exercise | Loss + Overall Weight | Loss + Monthly Weight + Exercise
Started | 4 (5 participants were not started with the intervention with this condition, because 1 participant was immediately withdrawn (without orientation to the condition) because of a staff member's error in assessing this participant's age eligibility) | 5 | 5 | 5 | 5 | 5 | 5 | 5
Completed | 3 | 4 | 4 | 5 | 5 | 4 | 5 | 5
Not Completed | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lottery + Monthly Weight | Lottery + Overall Weight + Exercise | Lottery + Overall Weight | Lottery + Monthly Weight + Exercise | Loss + Monthly Weight | Loss + Overall Weight + Exercise | Loss + Overall Weight | Loss + Monthly Weight + Exercise | Total
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 39
Age, Continuous [Mean (Full Range); unit: years] | 24.5 [20 to 33] | 27.2 [20 to 31] | 29.6 [23 to 36] | 26.5 [22 to 33] | 25.6 [20 to 35] | 25.4 [20 to 30] | 29.2 [25 to 33] | 29.4 [21.0 to 40] | 29.1 [20 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 39
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 3 | 4 | 5 | 5 | 5 | 5 | 4 | 5 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 4 | 4 | 4 | 3 | 2 | 3 | 24
  White | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 10
  More than one race | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Body Mass Index category (proportion with overweight and obesity) [Count of Participants; unit: Participants] | 2 | 3 | 3 | 3 | 3 | 2 | 5 | 1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Intervention Satisfaction Observed From Follow-up Survey
Description: At 32 weeks gestation participants will be asked to offer insight into program acceptability in each condition, as well as satisfaction to the program in general by answering an internet-based survey, that was developed for this study (not a standardized scale). The investigators will examine participants' survey responses regarding participants' satisfaction of the program (items are scored on a scale from 1 to 5, with 5 being the most positive).
Time Frame: Up to 32 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lottery + Monthly Weight | Lottery + Overall Weight + Exercise | Lottery + Overall Weight | Lottery + Monthly Weight + Exercise | Loss + Monthly Weight | Loss + Overall Weight + Exercise | Loss + Overall Weight | Loss + Monthly Weight + Exercise
Number analyzed (Participants) | 3 | 4 | 4 | 5 | 5 | 4 | 5 | 5
units on a scale
  How much would you recommend using an e-scale for managing GWG to a friend? | 5 [5 to 5] | 4.25 [3 to 5] | 4.25 [2 to 5] | 5 [5 to 5] | 4.8 [4 to 5] | 4.75 [4 to 5] | 4.8 [4 to 5] | 4.8 [4 to 5]
  How much would you recommend using a fitness tracker for managing GWG to a friend? | 4.67 [4 to 5] | 3.5 [2 to 5] | 5 [5 to 5] | 5 [5 to 5] | 4.4 [2 to 5] | 4.25 [3 to 5] | 4.6 [4 to 5] | 4.4 [3 to 5]
  How much would you recommend setting a weight gain goal for managing GWG to a friend? | 4.67 [4 to 5] | 4.25 [3 to 5] | 4.5 [3 to 5] | 5 [5 to 5] | 4.4 [3 to 5] | 4.75 [4 to 5] | 4.8 [4 to 5] | 4.6 [4 to 5]
  How much would you recommend setting a physical activity goal for managing GWG to a friend? | 4 [3 to 5] | 4.25 [3 to 5] | 4.5 [3 to 5] | 5 [5 to 5] | 5 [5 to 5] | 4.25 [3 to 5] | 4.8 [4 to 5] | 4.8 [4 to 5]

2. Primary Outcome: Recruitment Yields Observed From Enrollment Survey
Description: The number of participants initially recruited for the study will be closely monitored.
Time Frame: Up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lottery + Monthly Weight | Lottery + Overall Weight + Exercise | Lottery + Overall Weight | Lottery + Monthly Weight + Exercise | Loss + Monthly Weight | Loss + Overall Weight + Exercise | Loss + Overall Weight | Loss + Monthly Weight + Exercise
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Participants | 4 | 5 | 5 | 5 | 5 | 5 | 5 | 5

3. Primary Outcome: Program Retention Observed From Enrollment and Followup Surveys
Description: The number of participants stayed in the study within the time frame of the study will be closely monitored.
Time Frame: Up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lottery + Monthly Weight | Lottery + Overall Weight + Exercise | Lottery + Overall Weight | Lottery + Monthly Weight + Exercise | Loss + Monthly Weight | Loss + Overall Weight + Exercise | Loss + Overall Weight | Loss + Monthly Weight + Exercise
Number analyzed (Participants) | 4 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Participants | 3 | 4 | 4 | 5 | 5 | 4 | 5 | 5

4. Secondary Outcome: Gestational Weight Gain Observed From Weight Recorded at Baseline and up to 36 Weeks
Description: At all measurement visits, weight will be recorded in kilograms on a calibrated research-grade scale. Weight will be measured on a calibrated digital scale in duplicate, with the participant wearing light clothing and no shoes. While we will obtain the mother's weight at baseline, we will also obtain self-reported preconception weight (before the last menstrual period). We will calculate the participant's GWG goal based on self-reported preconception BMI. The difficulty of anticipating when a final weight should be obtained to capture the fullest extent of GWG was considered, and we elected to use an approach that afforded two possible weights that would be available for analytic purposes. The Week 36 weight will be the primary outcome except for mothers who deliver prior to 36 weeks, in which case we will use the Week 32 weight.
Time Frame: Up to 36 weeks
Measure: Mean (Full Range); unit: kilograms gained
Arm/Group | Lottery + Monthly Weight | Lottery + Overall Weight + Exercise | Lottery + Overall Weight | Lottery + Monthly Weight + Exercise | Loss + Monthly Weight | Loss + Overall Weight + Exercise | Loss + Overall Weight | Loss + Monthly Weight + Exercise
Number analyzed (Participants) | 3 | 4 | 4 | 5 | 5 | 4 | 5 | 5
kilograms gained | 13.2 [10.0 to 18.0] | 6.8 [0.9 to 11.2] | 8.4 [-3.7 to 14.2] | 9.4 [8.1 to 11.2] | 9.6 [-2.1 to 20.1] | 8.9 [-0.2 to 13.3] | 11.8 [3.4 to 18.8] | 11.8 [6.9 to 15.0]

5. Secondary Outcome: Number of Participants With Gestational Weight Gain Within IOM Recommendation
Description: We will evaluate whether participants' final gestational weight gain at Week 32 or Week 36 pregnancy would be under, within, or above IOM's recommendation. The Week 36 weight will be the primary outcome except for mothers who deliver prior to 36 weeks, in which case we will use the Week 32 weight. This is to determine the effect of the intervention on prevention of excess gestational weight gain.
Time Frame: Up to 36 weeks pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | Lottery + Monthly Weight | Lottery + Overall Weight + Exercise | Lottery + Overall Weight | Lottery + Monthly Weight + Exercise | Loss + Monthly Weight | Loss + Overall Weight + Exercise | Loss + Overall Weight | Loss + Monthly Weight + Exercise
Number analyzed (Participants) | 3 | 4 | 4 | 5 | 5 | 4 | 5 | 5
Participants | 2 | 2 | 0 | 1 | 2 | 2 | 1 | 3

ADVERSE EVENTS:
Time Frame: Baseline to 36 weeks gestation
Description: Data on adverse events, consistent with the clinicaltrials.gov definition, were collected at data collection visits and as reported by participants in the interim
Arm/Group | Lottery + Monthly Weight | Lottery + Overall Weight + Exercise | Lottery + Overall Weight | Lottery + Monthly Weight + Exercise | Loss + Monthly Weight | Loss + Overall Weight + Exercise | Loss + Overall Weight | Loss + Monthly Weight + Exercise
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/5 | 1/5 | 1/5 | 0/5 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lottery + Monthly Weight (N=4) | Lottery + Overall Weight + Exercise (N=5) | Lottery + Overall Weight (N=5) | Lottery + Monthly Weight + Exercise (N=5) | Loss + Monthly Weight (N=5) | Loss + Overall Weight + Exercise (N=5) | Loss + Overall Weight (N=5) | Loss + Monthly Weight + Exercise (N=5)
Premature birth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 (0)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT03834194/Prot_SAP_000.pdf